CLINICAL TRIAL: NCT05993754
Title: Impact of Non-pharmacological Measures Applied by the Nursing Team in Reducing the Incidence of Postoperative Delirium During the Postoperative and 24hr After Surgery in Frail Elderly Undergoing Elective Non-cardiac Surgeries.
Brief Title: Non-pharmacological Prevention of POD in Frailty Elderly Undergoing Elective Surgery Applied by Nursing Teams
Acronym: NPPOD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 220727001
Record Dates: First submitted 2023-07-27; First posted 2023-08-15 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Frail Elderly Syndrome; Primary Prevention; Postoperative Delirium; Frailty
Keywords: Delirium; Non-pharmacological; Elderly; Frailty; Nursing; Postoperative
MeSH Terms: conditions — Emergence Delirium; Frailty; Delirium

STUDY DESIGN:
Intervention Model Description: Control group and intervention group
Who Masked: Participant, Care Provider
Masking Description: After signed informed consent at the preoperative unit and during the post anesthesia unit care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Frail and pre-frail elderly people over 65 years of age who underwent elective non-cardiac surgeries who receive non-pharmacological interventions by the nursing team
  Interventions: Other: Non-pharmacological intervention
- Control group (No Intervention): Frail and pre-frail elderly people over 65 years of age undergoing elective non-cardiac surgeries who will receive traditional care.

INTERVENTIONS:
Other: Non-pharmacological intervention — The intervention consists of six main elements:
  Correction of sensory deficits: Before surgery, the use of glasses, hearing aids and/or removable dental prostheses will be allowed, which will be removed before starting anesthesia in the emergency room. After surgery, they will be delivered back to the user.
  Reorientation: In the postoperative period, the person will be informed where they are and the visit of the companion will be coordinated.
  Early mobilization: A protocolized mobilization routine will be applied according to pain, state of consciousness, risk of thromboembolic disease and risk of falls.
  Environmental management: You will be shown the time on a clock, it will reinforce the idea of the place where you are and that you can count on the team in case you need assistance.
  Sleep protocol: The elderly person who does not want or cannot perform the mobilization routine, non-pharmacological sleep will be privileged.
  Reduction of anticholinergic drugs
  Arms: Intervention group

SUMMARY:
The increase in the population over 60 years of age who could receive surgery due to changes in life expectancy and advances in surgical and anesthetic techniques.

Likewise, elderly people (EP) may have a higher risk of postoperative morbidity and mortality compared to young people, with frailty being one of the risk factors that increases adverse outcomes in this period and increases the probability of developing syndromes such as postoperative delirium (POD).

Assessment of frailty in EP prior to surgery is not routine, so it is unknown how many frail and/or pre-frail EP undergo surgery in health care systems. There is an association between being frail and developing greater delirium and/or postoperative cognitive deficit, which in summary translates into an increase in perioperative morbidity and mortality.

For the prevention of POD, there are pharmacological and non-pharmacological measures that seek to promote orientation with respect to their environment and make it as familiar as possible, stimulate early aspects of memory and thinking skills, as well as promote sleep using environmental hygiene measures.

In Chile, protocols of non-pharmacological measures have been proposed by occupational therapy teams, which have had positive results in reducing POD in frail elderly patients. These measures are temporal-spatial reorientation, physical mobilization, correction of sensory deficits, environmental management, sleep protocol, and reduction of anticholinergic drugs with statistically significant results in the reduction of POD.

In accordance with the above, the objective of this study is to evaluate the impact of non-pharmacological measures applied by the nursing team in reducing the incidence of POD during the post-surgical period in fragile and pre-fragile EP undergoing elective non-cardiac surgeries.

It is expected that in the end, frail and pre-frail EP who receive non-pharmacological interventions by the nursing team will present a lower incidence of POD at 24 hours compared to those who receive traditional care.

DETAILED DESCRIPTION:
Participants will correspond to frail and pre-frail people over 65 years of age who undergo elective non-cardiac surgery that requires general anesthesia and who attend the UC-Christus Clinical Hospital.

Frailty instruments (FRAIL scale) and Clinical Frailty Scale (CFS) will be applied, together with a preoperative cognition test (MiniCog; in case of presenting an altered result, the Montreal Cognitive Assessment, MoCA instrument will be applied), the delirium screening test (Delirium Triage Screen, DTS; in case of presenting an altered result, the Confusion Assessment Method instrument will be applied. d, CAM). Then, the participants will be randomized into two groups:

1. A first group to which a protocol of non-pharmacological interventions implemented by the nursing team will be applied to prevent post-surgical delirium
2. A second control group that will only receive traditional care. The users of the first group who use glasses, hearing aids and/or removable dental prostheses will move from the pre-operative unit room to the surgical ward with these elements, which will be delivered to their caregiver or companion after the safety break and before starting anesthesia inside the ward room where they will be operated on.

Both groups will undergo standard monitoring (ECG, NIBP, SatO2) and anesthesia will be guided using frontal EEG (SedLine or bilateral BIS). During the intraoperative period, an effort will be made to maintain a Mean Blood Pressure ± 20% of baseline and to keep the patient normothermic.

In the postoperative stage, therapeutic activities of cognitive stimulation and socialization will be carried out where temporal-spatial information will be delivered, the visit of the companion will be coordinated, a protocolized mobilization routine will be carried out considering pain, state of consciousness, thromboembolic risk and risk of falls. In the event that she does not want or cannot carry out the protocolized mobilization routine, non-pharmacological sleep will be privileged.

One hour after the patient's admission to the recovery unit, a delirium evaluation will be performed using CAM by personnel other than the one who performed the non-pharmacological measures. Two hours later, the non-pharmacological measures will be reinforced and later a new evaluation of delirium will be applied using CAM.

An evaluation of delirium will be carried out during the morning by means of CAM 24 hours after the admission of the patient to the recovery unit by a person other than the nursing team, who has not applied the protocol of non-pharmacological measures.

If the elderly person is still hospitalized, a final delirium evaluation will be carried out by means of CAM during the afternoon (24 hours after admission to the recovery unit).

In the event that the person presents CAM (+), the application of non-pharmacological measures will be evaluated with the treating team and the respective interconsultation will be processed with the geriatric team of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 65 years
* Elective non-cardiac surgery
* General anesthesia with Bilateral BIS electroencephalographic monitoring or SedLine
* ASA I, II or III.

Exclusion Criteria:

* Neurosurgical patients
* History of alcohol and/or drug abuse
* History of recreational psychoactive drug use
* Allergy to anesthetic drugs.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirum (POD) | : 10 minutes, 60 minutes, 120 minutes, 720 minutes and 1440 minutes after anesthesia
  Neurocognitive syndrome can occur from anywhere after anesthesia measure using the Confusion assessment method (CAM). For a diagnosis of delirium by CAM, the patient must display presence of acute onset and fluctuating discourse and Inattention, and either disorganized thinking or Altered level of consciousness (positive CAM), otherwise, the result is negative (negative CAM).

SECONDARY OUTCOMES:
Frailty _FRAIL | Pre Anesthesia period at same day of the surgery
  Frailty elderly measure by FRAIL Scale. It assesses 5 components: fatigue, resistance, ambulation, illnesses, and loss of weight. The score goes from 0 to 5 and represents the state of health and each component is worth 1 point, where it is recorded as robust (0), pre-frail (1-2) and fragile (3-5).
Frailty_CFS | Pre Anesthesia period at same day of the surgery
  Frailty elderly measure by Clinical Frailty Scale (CFS). Present a score from 1 (very fit) to 9 (terminally ill) is given based on the descriptions and pictographs of activity and functional status.
Screening of Cognitive impairment_MiniCog | Pre Anesthesia period at same day of the surgery
  Using Mini-Cog Score: 0 to 2 indicates possible cognitive disorder; 3 to 5 indicates no cognitive disorder.
Possible Cognitive impairment_MoCA | Pre Anesthesia period at same day of the surgery
  Measure by Montreal Cognitive Assessment (MoCA) test The cut-off point for MCI-a is <21 and for mild dementia <20. If the person has less than 12 years of schooling, 1 point is added.
Risk of anesthesia | Pre Anesthesia period at same day of the surgery
  Using the American Society of Anesthesiologists (ASA) classification. Categorize the patient's risk of undergoing any procedure that requires anesthesia, allowing to assess their physiological state and systemic diseases. The ASA score is based on five classes (I to V).
  I. Patient is a completely healthy fit patient. II. Patient has mild systemic disease. III. Patient has severe systemic disease that is not incapacitating. IV. Patient has incapacitating disease that is a constant threat to life. V. A moribund patient who is not expected to live 24 hour with or without surgery.
Type of surgery | Pre Anesthesia period at same day of the surgery
  Classification of surgery by specialty
Educational level of chile | Pre Anesthesia period at same day of the surgery
  Using the number of years of formal learning
Type of Anesthesia | Up to 30 minutes after the end of the surgery
  Classification type of anesthesia (Total Intravenous anesthesia, Total inhalation anesthesia and/or other)
Electroencephalogram monitoring during the anesthesia | Up to 30 minutes after the end of the surgery
  Measure by electroencephalogram (EEG) monitor (SedLine or BIS). From the start of anesthesia to the end of it.
Type of drugs during anesthesia | Up to 30 minutes after the end of the surgery
  According of classification type of anesthesia, amount of total drugs (mg, mcg, %etgas and/or other) General anesthesia (gas-based anesthesia or total intravenous anesthesia)
Postoperative Pain | 10 minutes, 60 minutes, 120 minutes, 720 minutes and 1440 minutes after anesthesia
  Measure by Numerical Rating Scale (NRS) pain The patient indicates the degree of pain on a scale of 0-10, where 0 is no pain and 10 is the worst pain imaginable.
Positive POD Positive CAM: presence of post-operative delirium (POD) Negative CAM:. absence of postoperative delirium (POD) | 720 minutes and 1440 minutes after anesthesia
  Measure by type of pharmacological measure by type of pharmacological management

CONTACTS AND LOCATIONS:
Overall Officials: Victor Contreras, MSN, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile